CLINICAL TRIAL: NCT04377347
Title: Time From First Health Care Contact to Neurosurgical Admission and the Effect on Long-term Labour Market Affiliation and Mortality in Patients With Spontaneous Subarachnoid Haemorrhage
Brief Title: Long-term Effects of Time to Treatment in Subarachnoid Haemorrhage
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Asger Sonne, MD, Principal investigator, Rigshospitalet, Denmark
Other Study IDs: Outcome
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Time

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Confirmed spontaneous subarachnoid haemorrhage: Patients, minimum 18 years of age, identified with the diagnosis in the Danish National Patient Register. The diagnosis is verified by medical record review.
  All patients were initially admitted to a hospital in the Capital Region of Denmark.
  In a national labour marked register and the civil registration register the patients are then followed for four years.
  Interventions: Other: Time

INTERVENTIONS:
Other: Time — Exposure is the time from patients call the Emergency Medical Coordination Center to they are admitted to a neurosurgiocal department.

SUMMARY:
For patients with spontaneous subarachnoid haemorrhage, it remains to be investigated if there is an association between the time from patients call the Emergence Medical Coordination Center to neurosurgical admission and long-term outcome.

This is a retrospective cohort study with four-year followup. The primary aim is to determine if the time to neurosurgical admission is associated to labour marked affiliation and mortality after four years.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous subarachnoid haemorrhage registered in the Danish National Patient Register and confirmed by medical record review.
* Initially admitted to a hospital in the Capital Region of Denmark between 1 January 2008 and 31 December 2014.

Exclusion Criteria:

* Prior subarachnoid haemorrhage.
* Inhospital symptom onset.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are retired or on social transfer payments the last three months before the sSAH are excluded from analyses on retirement and labour marked affiliation. However, they are included in mortality analyses. Also, patients aged 60 years or older are excluded in analyses of early retirement as reduced work capacity may to a higher degree result in early voluntary retirement.
Sampling Method: Non-Probability Sample
Enrollment: 537 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Labour marked affiliation and mortality | 4 years
  The incidence of all-cause death and early retirement over the four-years after sSAH for different times to treatment is shown with Kaplan-Meier plots, and assessed with log-rank tests.

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No